CLINICAL TRIAL: NCT07277933
Title: Efficacy and Safety of KHN702 Tablets in Moderate to Severe Post-operative Pain Patients: A Randomized, Double-blind, Placebo-Controlled, Phase Ib Trial
Brief Title: Efficacy and Safety of KHN702 Tablets in Moderate to Severe Post-operative Pain Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Kanghong Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KHN702-30102
Record Dates: First submitted 2025-11-28; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KHN702 (Experimental): Participants will be randomized to either the KHN702 tablet or placebo group, and administer study drug for 2 days.
  Interventions: Drug: KHN702
- KHN702 placebo (Placebo Comparator): Participants will be randomized to either the KHN702 tablet or placebo group, and administer study drug for 2 days.
  Interventions: Drug: KHN702 placebo

INTERVENTIONS:
Drug: KHN702 — KHN702 tablet for oral administration
  Arms: KHN702
Drug: KHN702 placebo — KHN702 placebo tablet for oral administration
  Arms: KHN702 placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, parallel-group clinical trial. To preliminarily evaluate the safety and efficacy of KHN702 tablets in moderate to severe post-operative pain patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between the ages of 18 and 75 years, inclusive.
2. Body mass index (BMI) of 18.0 to 30.0 kg/m2, inclusive.
3. Patients scheduled for surgery.
4. According to the researcher's medical judgment, American Society of Anesthesiologists (ASA) classification≤Grade II.
5. The subject can understand and comply with the study procedures and requirements, and can provide written informed consent prior to any study procedures.
6. NRS ≥ 4 points within 6 hours after surgery.

Exclusion Criteria:

1. Participants experiencing acute or chronic pain unrelated to the surgical site, which the investigator deems may confound the participant's assessment of postoperative pain.
2. History or evidence of any of the following conditions prior to screening:

   * History of significant cardiovascular or cerebrovascular disease;
   * Severe respiratory disease history;
   * Severe Neurological and Psychiatric disease History;
   * Active peptic ulcer disease, significant vomiting, chronic diarrhea, ileus, malabsorption, or other known conditions that significantly affect drug absorption, distribution, metabolism, or excretion;
   * Subjects at high risk of bleeding who are deemed unsuitable for this trial by the investigator;
3. Long-term use of opioids or nonsteroidal anti-inflammatory drugs within the past 30 days prior to screening, or discontinuation of medications affecting analgesic efficacy assessment (except those permitted by the protocol) less than 5 half-life prior to randomization.
4. Subjects with a history of opioid allergy, or those with a history of allergy to the intraoperative medications specified in the protocol, postoperative rescue analgesics, or known allergies to the investigational drug or its excipients.
5. Subjects who underwent major surgery within 3 months prior to screening and the investigator determined that it would affect postoperative pain assessment.
6. Any of the following infectious diseases were present during screening: Hepatitis B surface antigen (HBsAg) positive, hepatitis C virus antibody (HCV Ab) positive, human immunodeficiency virus antibody (HIV Ab) positive, or serum treponema pallidum antibody (TPAb) positive.
7. History of substance abuse or alcohol abuse within the three months prior to screening .
8. History of blood donation within the past three months prior to screening.
9. Individuals who have participated in any clinical research within the past three months prior to screening .
10. Pregnant or lactating women; women or men of reproductive potential who are unwilling to use contraception throughout the study period; or subjects (including male subjects) planning to conceive within 3 months after study completion.
11. Subjects with intraoperative blood loss exceeding 1000 mL or those experiencing other severe complications during surgery;
12. Subjects requiring intensive care following surgery;
13. Other circumstances deemed unsuitable for participation in this trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Time-weighted the Sum of Pain Intensity Differences in Pain Score 0 to 48 hours after the first dose | 48 hours

SECONDARY OUTCOMES:
Safety：Incidence and severity of Adverse Events( AE)/SAE | from ICF signing date to day 7 since the first dose
Cmax | 48 hours
  Maximum Plasma Concentration
Time-weighted the Sum of Pain Intensity Differences in Pain Score over Times | 48 hours
Times and Cumulative Amount of Rescue Analgesics Used by Subjects within 0 to 48 Hours after the First Dose. | 48 hours
Tmax | 48 hours
  Time to Maximum Plasma Concentration
AUC0-t | 48 hours
  Area Under the concentration-time curve from zero to t

IPD SHARING:
Plan to Share IPD: Undecided